CLINICAL TRIAL: NCT06823336
Title: The SHINE (Supporting Her In Navigating Exercise) Program: A Pilot Study Examining Peer Support as an Exercise Promotion Tool Among Undergraduate Women Initiates
Brief Title: The Supporting Her In Navigating Exercise Program: Examining Peer Support to Promote Exercise Among Undergraduate Women
Acronym: SHINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); St. Joseph's Care Group (Other)
Responsible Party: Principal Investigator, Erin Pearson, Associate Professor, Lakehead University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 195012
Record Dates: First submitted 2025-01-28; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Social Support (Formal and Informal)
Keywords: Exercise psychology; Peer-mentorship program; Womens health; Pandemic recovery era; mixed methods; Undergraduate women
MeSH Terms: interventions — Methods; Exercise

STUDY DESIGN:
Intervention Model Description: This study will include two conditions: an intervention (exercise plus mentor) and a control (exercise only) condition. Both groups will be encouraged to engage in exercise at least three times a week for 30 minutes at the campus facilities for 6-weeks. The intervention group will additionally engage in one-on-one exercise at the campus facilities once a week with their randomly assigned peer mentor and virtually communicate between sessions. Thus, intervention participants will be engaging in independent exercise at least twice a week. Those assigned to the control condition will only engage in independent exercise at least three times a week.
Who Masked: Investigator
Masking Description: The student researcher will be masked to the two conditions during the participant's orientation session (e.g., facility tour, baseline data collection) and will only reveal their condition using a numbered opaque sealed envelope immediately following data collection. The participant will be asked to hold this allocation in confidence and initiative contact with their mentor to schedule the first workout session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise plus mentor (Experimental): Participants will be encouraged to engage in independent exercise twice a week for 30 minutes. They will be randomly assigned to a peer-mentor, with whom they will engage in on-on-one exercise once a week for 30 minutes. Between sessions, they will engage in virtual communication with each other for about 30 minutes each week. Each participant-mentor duo will continue this protocol for 6-weeks.
  Interventions: Other: Intervention
- Exercise alone (Active Comparator): Participants will be encouraged to engage in exercise three times a week for thirty minutes, over a span of 6-weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — Participants will be encouraged to engage in independent exercise twice a week for 30 minutes. They will be randomly assigned to a peer-mentor, with whom they will engage in on-on-one exercise once a week for 30 minutes. Between sessions, they will engage in virtual communication with each other for about 30 minutes each week. Each participant-mentor duo will continue this protocol for 6-weeks.
  Other Names: Social support
  Arms: Exercise plus mentor
Other: Control — Participants will be encouraged to engage in exercise three times a week for thirty minutes, over a span of 6-weeks.
  Other Names: Exercise alone
  Arms: Exercise alone

SUMMARY:
The purpose of this randomized controlled pilot trial is to test the effectiveness of a six-week tailored physical activity program with and without peer mentoring on the psychological constructs and exercise behaviour of inactive undergraduate women. The objectives are to:

* Quantify the degree to which a peer-mentorship intervention affects exercise motivation determined through three basic psychological needs (i.e., autonomy, competence, and relatedness).
* Examine general psychological distress and exercise engagement throughout the study.
* Qualitatively explore participants' experiences following the completion of the program using an open-ended survey to gain a better understanding of its impact.

Researchers will compare the parallel arm conditions to see how the inclusion of social support impacts exercise engagement.

Participants will be asked to engage in exercise three times a week at the campus gym; those in the intervention condition will have an assigned peer-mentor who will join them for one weekly session and virtually communicate with them between sessions.

DETAILED DESCRIPTION:
This study aims to explore the use of social support as an exercise promotion tool among undergraduate women who don't exercise or who do so occasionally.

Senior undergraduate and graduate women at Lakehead University were recruited as study mentors for this research project. These individuals were required to have a health background with expertise in physical activity, engage in 150 minutes of exercise per week, be familiar with the university's fitness facility, and be willing to help others become more active. Once confirmed, mentors were trained via a two-hour workshop, focusing on program roles and responsibilities, motivational strategies, physical activity structuring, and communication/confidentiality guidelines.

For participants to be considered eligible, they need to engage in , once deemed eligible via an eligibility questionnaire, all participants will engage in a baseline orientation session. During this session, they will meet with the student researcher in a private room in the C.J. Sanders Fieldhouse at Lakehead University. During this meeting, the duo will review the information letter/participant rights, and if in agreement, the participant will provide informed consent. Once this occurs, the participant will complete a baseline survey that includes a number of measures (e.g., demographic questions, Depression Anxiety Stress Scale, Behavioural Regulation in Exercise Questionnaire, and Psychological Needs Satisfaction in Exercise Questionnaire), and have their height and weight recorded. They will then create a confidential Strava account, to enable exercise tracking and friend the SHINE Program account. Following this, participants will receive a facility tour, where the student researcher will show them around the campus fitness facility and demonstrate how to use some equipment in each space. Once the facility tour is completed, the student researcher will select a sequentially numbered opaque envelope sealed by the research team, indicating which condition the participant will be assigned to. Participants assigned to the exercise condition will be invited to ask questions as their orientation has concluded, while intervention participants will review communication guidelines, create a GroupMe account, and be assigned to a mentor based on mutual availability.

All participants in this study will be asked to engage in exercise three times a week for 30 minutes at the campus gym facility. Individuals assigned to the intervention condition will be joined by their peer-mentor in one of these sessions once a week and be asked to engage in virtual communications in between sessions.

This will continue for 6-weeks, with additional data collection occurring at weeks 3 and 6. Upon completion of the study at week 6, participants will be asked to complete an open-ended exit questionnaire to explore their program experiences.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a woman
* Full-time undergraduate student at Lakehead University
* Classified as an exercise initiate (e.g., report one or fewer bouts of exercise per week)
* Reported an absence of health risks that would interfere with exercise engagement as determined by the Get Active Questionnaire
* Able to commute to Lakehead's campus
* Want to become more active
* Have access to online technology (e.g., email, zoom)
* Can speak, read, and write in English fluently

Exclusion Criteria:

* Identify as a man
* Not enrolled as a full-time undergraduate student at Lakehead University
* Report the presence of health risks that would interfere with exercise engagement
* Meet the national physical activity guidelines (e.g., 150 minutes of moderate to vigorous exercise per week)
* Unable to commute to campus
* Lack of access to technology
* Not fluent in English

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Girls/women have historically engaged in less exercise than those of boys/men at all ages, a trend that largely worsens in young adulthood. Post-removal of pandemic precautions, the exercise habits of undergraduate women disproportionately decreased as compared to those of men. Thus, a need to focus on this population and provide them with a gender specific exercise program to meet their unique needs exists.
Enrollment: 24 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Psychological Needs Satisfaction in Exercsie Scale | During enrollment at baseline, after week 3, and at the end of the study at week 6
  Participants' exercise motivation, focused on the psychological needs and specific regulations, will be assessed quantitatively using The Psychological Needs Satisfaction in Exercise Scale. This 18-question tool, participants will evaluate each statement based on how it applied to them over the past week on a six-point scale (1= false, 6= true). In this scale, six statements are allotted for each of the three basic needs (e.g., autonomy, competence, and relatedness) in the context of exercise engagement. Subscale scores will be calculated by averaging the six items assigned to each basic psychological need, with higher scores being more indicative of greater self-determination and lower of less.
Behavioural Regulation in Exercise Questionnaire- 3 | During enrollment at baseline, after week 3, and at the end of the study at week 6
  This questionnaire will be used to to gauge where an individual falls on the six-point motivational continuum, as it relates to exercise engagement. This will be assessed quantitatively using the Behavioural Regulation in Exercise Questionnaire-3, as participants will evaluate each statement based on how it applied to them over the past week. The 24-questions in this measure operate on a five-point Likert scale (0= not true for me, 2= sometimes true for me, 4= very true for me). In this questionnaire, four statements have been allocated for each of the six types of regulation/motivation (e.g., motivation, introjected regulation, identified regulation, integrated regulation, intrinsic regulation, external regulation). Subscale scores will be calculated by averaging the six items assigned to each basic psychological need, with higher scores being more indicative of greater intrinsic motivation and lower of greater extrinsic motivation.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale- Short Form | During enrollment at baseline, following week 3, and at the end of the study at week 6
  Participants' general psychological distress will be quantitatively measured through the Depression Anxiety Stress Scale- Short Form. The 21-question scale operates on a four-point Likert scale (0= never, 1= sometimes, 2= often, 3= almost always), and asks participants to evaluate each statement based on how it applied to them over the past week. In this scale, seven questions were allotted to each of the three categories (e.g., depression, anxiety, and stress). When scoring the DASS-21, the scores for each of the three categories are independently summed to gain a final score, with higher scores being indicative of severe psychological distress and lower scores suggest average or typical symptoms.
Exercise Tracking- Gym location | From enrollment to the end of the program at 6 weeks
  Participants' exercise engagement will be measured via a virtual exercise monitoring platform, Strava. Participants will upload their workouts each week, revealing the area of the gym they used (e.g., Hangar, Wolf Den, Basement).
Exercise Tracking- Duration | From enrollment to the end of the program at 6 weeks
  Participants' exercise engagement will be measured via a virtual exercise monitoring platform, Strava. Participants will upload their workouts each week, revealing the duration of their session.
Exercise Tracking- Workout Details | From enrollment to the end of the program at 6 weeks
  Participants' exercise engagement will be measured via a virtual exercise monitoring platform, Strava. Participants will upload their workouts each week, revealing the type of workout they engaged in (e.g., cardio, upper body strength, lower body strength, full body strength training).
Exercise Tracking- Frequency | From enrollment to the end of the program at 6 weeks
  Participants' exercise engagement will be measured via a virtual exercise monitoring platform, Strava. Participants will upload their workouts each week, revealing the number of sessions they engage in each week.

OTHER OUTCOMES:
Qualitative Experiential Accounts- Open Ended Questionnaire | Findings will be collected upon completion of the program, at the end of week 6.
  Upon completion of the program, all participants will complete an open-ended questionnaire to gain an in-depth understanding of their program experiences. This questionnaire is comprised of open-ended questions adopted from previous research in this area and includes questions regarding topics such as exercise habits, motivation, three basic psychological needs, and perceptions of the SHINE program.
Facility Usage Data- Frequency | From enrollment to the end of the program at 6 weeks
  Facility usage data will be monitored through Lakehead University's Athletics platform and will include dates and times signed in at the gym.
Communication Data- Frequency | From enrollment to the end of the program at 6 weeks
  Communication usage data between participants and their peer mentors will be monitored by the student researcher through GroupMe, an online messaging platform.
Demographic Information- Program of study | During enrollment at baseline
  Demographic questions to assist the researchers in understanding the population characteristics will be asked at the outset of the study, including their program of study.
Demographic Information- Year of study | During enrollment at baseline
  Demographic questions to assist the researchers in understanding the population characteristics will be asked at the outset of the study, including the year of study they are currently completing in their program.
Demographic Information- Birth country | During enrollment at baseline
  Demographic questions to assist the researchers in understanding the population characteristics will be asked at the outset of the study, including their birth country.
Demographic Information- Ethnicity | During enrollment at baseline
  Demographic questions to assist the researchers in understanding the population characteristics will be asked at the outset of the study, including their ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Erin S Pearson, PhD, Principal Investigator — Lakehead University
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
No decision has been made thus far. The research team will decide once the data collection period is completed, based on the number of participants who complete the study.

REFERENCES:
- [Background] DeShaw KJ, Lansing JE, Perez ML, Ellingson LD, Welk GJ. Effects of a peer health coaching program on college student lifestyle behaviors. J Am Coll Health. 2024 Dec;72(9):3330-3337. doi: 10.1080/07448481.2022.2155473. Epub 2023 Jan 3. PMID 36595662
- [Background] Keeler, L. A., Skidmore, B., Leenstra, T., MacDonald, J. R., & Stewart, D. (2021). Treating university students' depression using physical activity with peers: Two field-based quasi-experiments grounded in the self-determination theory. Journal of College Student Psychotherapy, 35(3), 205-223. https://doi.org/10.1080/87568225.2019.1660293